CLINICAL TRIAL: NCT04636489
Title: An Interventional Study for the Effects of Highland Barley β-glucan on the Management of Glucose Metabolism and Insulin Sensitivity
Brief Title: Effect of Prebiotics on Blood Glucose Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Min Xia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020HBβG-D
Record Dates: First submitted 2020-11-18; First posted 2020-11-19 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Hyperglycemia; Insulin Sensitivity
Keywords: Hyperglycemia; Prebiotics
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: placebo-controlled, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and care providers at the scene are all blinded to the allocation of treatment group. Data collected will be analyzed by another investigator who is blinded to the study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Highland barley β-glucan group (Experimental): Participants will be given oral liquids mainly containing highland barley β-glucan once daily for 8 weeks followed by comprehensive physical and clinical examinations.
  Interventions: Dietary Supplement: Highland barley β-glucan dietary supplement
- Placebo group (Placebo Comparator): Participants will be given oral liquids mainly containing Corn starch once daily for 8 weeks followed by comprehensive physical and clinical examinations.
  Interventions: Other: Placebo controls

INTERVENTIONS:
Dietary Supplement: Highland barley β-glucan dietary supplement — 100 mL oral liquid mainly containing highland barley β-glucan once daily for 8 weeks
  Arms: Highland barley β-glucan group
Other: Placebo controls — Placebo with a similar appearance and taste to highland barley β-glucan supplement
  Arms: Placebo group

SUMMARY:
This survey is designed to investigate the effect of highland barley β-glucan supplementation on the regulatory of blood glucose, gut microbiota and cardiovascular risk fators in subjects with hyperglycemia.

DETAILED DESCRIPTION:
Highland barley β-glucan belongs to the group of prebiotics and has been found to be associated with multiple health benefits. However, its protective role in subjects with hyperglycemia are remain unclear. This study aims to examine the effect of 8-week prebiotics supplementation on glucose management in subjects with hyperglycemia. By understanding the mechanism by which prebiotics exert the beneficial effects, we can better control the rising prevalence of hyperglycemia, which is a major risk factor for cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 30-65 years old
2. Fasting venous plasma glucose ≥5.6mmol/L OR plasma glucose 2 h after an oral glucose load ≥7.8mmol/L OR glycosylated hemoglobin ≥5.7% OR newly diagnosed diabetes without hypoglycemic drugs using
3. BMI≥18 kg/ m2

Exclusion Criteria:

1. Receiving or have been treated with hypoglycemic drugs or insulin.
2. Complications including cardiovascular and cerebrovascular diseases such as coronary heart disease and stroke.
3. Severe liver or renal insufficiency (alanine aminotransferase, aspartate aminotransferase or alkaline phosphatase is greater than 3 times the upper limit of normal OR GFR<30ml/min/1.73m2).
4. Autoimmune diseases or thyroid diseases.
5. Women who are pregnant, nursing, or prepare to give birth during the trail.
6. Malignant disease, infectious disease, inflammatory disease and advanced liver disease.
7. Mental or intellectual abnormalities, unable to sign informed consent.
8. Complications including chronic gastrointestinal disease; or suffered from acute gastrointestinal diseases within 1 months before screening visit.
9. Received antibiotics, probiotics within 3 months before screening visit or throughout the trail.
10. Major operations were performed within six months of screening visit, or will be made during the trial.
11. Alcohol abuse (alcohol intake>60g/d for male and alcohol intake>40g/d for female)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
fasting venous plasma glucose | baseline and after 8-week intervention
  changes of fasting venous plasma glucose levels
plasma glucose 2 h after an oral glucose load | baseline and after 8-week intervention
  changes of plasma glucose levels 2 h after an oral glucose load
glycosylated hemoglobin | baseline and after 8-week intervention
  changes of glycosylated hemoglobin levels

SECONDARY OUTCOMES:
gut microbiota | baseline and after 8-week intervention
  changes of gut microbiota
microbial metabolites | baseline and after 8-week intervention
  changes of microbial metabolites by untargeted metabolomics
Matsuda index | baseline and after 8-week intervention
  changes of Matsuda index based on OGTT
flow-mediated dilation | baseline and after 8-week intervention
  changes of flow-mediated dilation by VICORDER Complete Vascular Laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Min Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No